CLINICAL TRIAL: NCT02720640
Title: Safety and Efficacy of the Alpha AMS Subretinal Implant for Partial Restoration of Vision in Visually Impaired Participants With Degenerative Retinal Disease
Brief Title: Safety and Efficacy of the Alpha AMS Subretinal Implant
Acronym: OX-RI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E/2015/0119
Record Dates: First submitted 2015-12-04; First posted 2016-03-28 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Visual Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implant 'on' vs implant 'off' (Experimental): Intra-individual comparison of implant 'on' vs implant 'off'
  Interventions: Device: Implant 'on' vs implant 'off'

INTERVENTIONS:
Device: Implant 'on' vs implant 'off' — Single group assignment
  Other Names: Alpha AMS; Retinal Implant Alpha AMS; Retinal implant; Bionic eye; Retinal prosthesis; Sub retinal chip

SUMMARY:
The aim of this single-centre study is to assess the safety and efficacy of the Retina Implant Alpha AMS (Retina Implant AG, Reutlingen, Germany) in participants with severe visual impairment secondary to outer retinal degeneration caused by retinitis pigmentosa (RP). The study is sponsored by the University of Oxford and funded by the National Institute for Health Research (UK).

DETAILED DESCRIPTION:
The specific research questions are, i) can the implant partially restore vision to an eye with no light perception and ii) what are the safety implications for the ocular and periorbital tissues of the implanted eye? In advanced RP the light detecting photoreceptor cells of the retina degenerate slowly over time, and may eventually lead to blindness. The subretinal implant replaces the degenerate photoreceptor layer and stimulates the residual overlying healthy retinal layers in response to a light stimulus. These signals are then carried on to the brain along the normal visual pathway. Investigators are seeking to recruit six participants who fulfill the eligibility criteria, which include advanced RP with no useful light perception vision in the eye to receive the implant. Participants must be aged between 18 and 70 years old, be highly motivated, and be well enough for a general anaesthetic. The eye must have also had cataract surgery. The project will be conducted at the Oxford Eye Hospital. Those participants selected to receive the implant will be followed for 12 months from the date of surgery. Between week 1 and month 12 there will be at least 7 outpatient clinic visits for a range of visual tests and eye assessments. After 12 months the trial will officially end, however investigators will continue to review all research participants in clinic as would be standard care for a patient with RP. The implant may be removed at any stage e.g. when it ceases to function or at the participant's request.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 to 70 years old.
* Hereditary retinal degeneration of the outer retinal layers i.e. photoreceptor rods & cones.
* Angiography shows retinal vessels adequately perfused, despite pathological RP condition.
* Severe visual impairment (at least monocular) i.e. visual functions insufficient for localization of objects, self-sustained navigation and orientation e.g. impaired light localization or worse.
* Ability to read normal print in earlier life, optically corrected (without magnifying glass).
* Able to participate in the study during the full time period of one year.
* Pseudophakic in the eye to receive the implant.
* Stable dose of current regular medication for at least four weeks prior to trial entry.
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial.
* Participant has clinically acceptable laboratory and ECG results as confirmed at - Screening Visit and upon review by consultant anaesthetist.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Period of appropriate visual functions < 12 years / lifetime.
* Optical coherence tomography (OCT) shows significant retina oedema &/or scar tissue within target region for implant.
* Retina detected as too thin to expect required functionality of inner retina as shown via OCT.
* Lack of inner-retinal function, as determined by Electrically Evoked Phosphenes (EEP).
* Heavy clumped pigmentation at posterior pole.
* Any other ophthalmologic disease with relevant effect upon visual function (e.g. glaucoma, optic neuropathies, trauma, diabetic retinopathy, retinal detachment).
* Amblyopia reported earlier in life for eye to be implanted.
* Systemic diseases that might imply considerable risks with regard to the surgical interventions and anesthesia (e.g. cardiovascular/ pulmonary diseases, significant metabolic diseases e.g. diabetes).
* Neurological and/or psychiatric diseases (e.g. Parkinson, epilepsy, depression).
* Hyperthyroidism or hypersensitivity to iodine.
* Hypersensitivity to fluorescent dye (fluorescence angiography).
* Women who are pregnant or nursing, or women of childbearing age who are not willing to use a medically acceptable means of birth control for the duration of the study, or women unwilling to perform a pregnancy test before entering the study.
* Participation in another interventional clinical trial within the past 12 weeks.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Alpha AMS retinal implant system used for activities of daily living tasks. | 12 months
  Activities of daily living are assessed with implant ON versus OFF via:
  • Activities of daily living tasks

SECONDARY OUTCOMES:
Efficacy of the Alpha AMS retinal implant system used for partial restoration of visual acuity. | 12 months
  Visual acuity or light-perception and/or object-recognition assessed with implant ON versus OFF via
  • Freiburg visual Acuity and Contrast Test (FrACT)
Efficacy of the Alpha AMS retinal implant system used for partial restoration of basic light detection.. | 12 months
  Visual acuity or light-perception and/or object-recognition assessed with implant ON versus OFF via:
  • Basic Light and Motion test (BaLM)
Efficacy of the Alpha AMS retinal implant system used for partial restoration of grating acuity. | 12 months
  Visual acuity or light-perception and/or object-recognition assessed with implant ON versus OFF via:
  • Basic Grating Acuity test (BaGA).
Safety of the Alpha AMS retinal implant. | 12 months
  The number of participant with Adverse Events and/or Serious Adverse Events, as defined by the Study Protocol, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MacLaren, DPhil FRCS, Principal Investigator — 1. Nuffield Laboratory of Ophthalmology, Department of Clinical Neurosciences, University of Oxford; 2. Oxford Eye Hospital, Oxford University Hospitals NHS Foundation Trust; 3. Moorfields Eye Hospital NHS Foundation Trust, London
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cehajic Kapetanovic J, Troelenberg N, Edwards TL, Xue K, Ramsden JD, Stett A, Zrenner E, MacLaren RE. Highest reported visual acuity after electronic retinal implantation. Acta Ophthalmol. 2020 Nov;98(7):736-740. doi: 10.1111/aos.14443. Epub 2020 Apr 28. PMID 32343050
- [Derived] Stingl K, Schippert R, Bartz-Schmidt KU, Besch D, Cottriall CL, Edwards TL, Gekeler F, Greppmaier U, Kiel K, Koitschev A, Kuhlewein L, MacLaren RE, Ramsden JD, Roider J, Rothermel A, Sachs H, Schroder GS, Tode J, Troelenberg N, Zrenner E. Interim Results of a Multicenter Trial with the New Electronic Subretinal Implant Alpha AMS in 15 Patients Blind from Inherited Retinal Degenerations. Front Neurosci. 2017 Aug 23;11:445. doi: 10.3389/fnins.2017.00445. eCollection 2017. PMID 28878616